CLINICAL TRIAL: NCT06354374
Title: Relationship Between Soft Tissue Volume, Dimensions and Tomographic Alveolar Ridge Classification System for Dental Implant Treatment.
Brief Title: Soft Tissue Volume, Dimensions and Tomographic Alveolar Ridge Classification System for Dental Implant Treatment.
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: British University In Egypt (Other)
Responsible Party: Principal Investigator, ahmed hamdy mahmoud, assistant lecturer, Ain Shams University
Other Study IDs: 24-026
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Soft Tissue Volume

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: volume survey — All subjects will receive oral hygiene instructions and, if needed. A dental cleaning of plaque and calculus. After calibration using digital photographs and digital intraoral scans, CBCT scans will be taken as a prerequisite for dental implant treatment protocol. one dentist who will not be involved in the screening phase will obtain all clinical parameters (gingival biotype, probing depth, gingival thickness, gingival width) to avoid any bias. After finishing data collection, a customized treatment plan for each patient will be performed and dental implant treatment will be completed for each patient.

SUMMARY:
Despite the importance of soft tissue dimensions for periodontal, restorative, implant, and orthodontic treatment, the current classifications of tomographic alveolar ridge topography lack the soft tissue component(Tolstunov, 2014). Therefore, the present study will be to evaluate the relationship between soft tissue volume and the dimensions & tomographic alveolar ridge classes as well as to incorporate the soft tissue volumetric evaluation in the classification system.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients in a healthy systemic condition who required comprehensive dental treatment.
2. Both genders with age group > 18 years old.
3. Patients should have at least a single missing tooth that requires dental implant placement.
4. Healing period of 3 months after extraction prior to surgical procedures.
5. CBCT scans will be obtained as a part of the comprehensive dental treatment.
6. Patients should approve to deliver a signature to a written consent after studying nature explanation.

Exclusion Criteria:

1. Patients with severe smoking habits >10 cig \ day.
2. Pregnant females, decisional impaired individuals, Prisoners, and handicapped patients.
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures.
4. Patients on any medication affecting the soft tissue health (e.g., amlodipine, Cyclosporine A, hydantoin)
5. Patients with infections either periodontally or periapically

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross sectional observational clinical study will include 350 patients that will be recruited from the outpatient clinic of the department of Oral Medicine, Periodontology, and Diagnosis, Faculty of Dentistry, The British University in Egypt.
  Demographic data of all patients will be collected. Patients will be clearly instructed about the purpose of this study and will give their consent by signing an informed consent.
  The study will be started after being accepted by the faculty of Dentistry, The British University in Egypt Research Ethics Committee. The study tracks the guidelines of the research ethical committee in line with the Helsinki Declaration of 1975.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the relationship between soft tissue volume & tomographic alveolar ridge classes | 3 months
  the relationship between soft tissue volume and tomographic alveolar ridge classes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hamdy, Al Shorouk City, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided